CLINICAL TRIAL: NCT05251220
Title: Efficacy and Safety of the Neodymium Laser in Treatment of Urogenital Tract Diseases in Women
Status: Completed | Type: Observational
Sponsor: 1st Federal Budgetary Healthcare Institution Volga District Medical Center (Other Government)
Responsible Party: Principal Investigator, Pauzina Olga Alexandrovna, Head of the Outpatient Department of the Volga District Medical Center of the FMBA of Russia, Principal Investigator, 1st Federal Budgetary Healthcare Institution Volga District Medical Center
Other Study IDs: 29.10№14
Record Dates: First submitted 2021-12-12; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Genitourinary Syndrome of Menopause; Pelvic Floor Dysfunction; Vulvar Lichen Sclerosus
Keywords: neodymium laser, GUMS, lichen sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus; Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 10 women with objectively confirmed vulvovaginal atrophy: 10 women with objectively confirmed vulvovaginal atrophy (genitourinary menopausal syndrome
- 37 women with 1-2 degree prolapse of the vaginal walls combined with stress urinary incontinence: 37 women with 1-2 degree prolapse of the vaginal walls combined with stress urinary incontinence
- 7 with vaginal relaxation syndrome: 7 with vaginal relaxation syndrome
- 6 with vulvar lichen sclerosus: 6 with vulvar lichen sclerosus

SUMMARY:
Study objective: To evaluate the efficacy and safety of the Magic Max neodymium laser in the medical treatment of women with symptoms of genitourinary syndrome of menopausal, vulvar lichen sclerosus and pelvic floor muscle reduction.

DETAILED DESCRIPTION:
Study objective: To evaluate the efficacy and safety of the Magic Max neodymium laser in the medical treatment of women with symptoms of genitourinary syndrome of menopausal, vulvar lichen sclerosus and pelvic floor muscle reduction.

Materials and methods: 60 patients with diseases of the urogenital tract were enrolled into the study; they were treated with a neodymium (ND) laser: three 20-minute sessions every 28 ± 2 days. Efficacy was assessed by means of the Female Sexual Function Index (FSFI), ICIQ-SF, PISQ-12, SF36 survey forms, and a questionnaire to identify urinary disorders at the following time points: before treatment, one month after each session and 6 months after the last procedure.

ELIGIBILITY:
Inclusion Criteria:

* diseases of the urogenital tract
* symptoms of genitourinary menopausal syndrome,
* vulvar lichen sclerosus
* pelvic floor muscle reduction

Exclusion criteria:

* pregnancy
* oncological diseases

Ages: 29 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patients with diseases of the urogenital tract were enrolled into the study;women with symptoms of genitourinary menopausal syndrome, vulvar lichen sclerosus and pelvic floor muscle reduction
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Change in vaginal dryness from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by SF36 quality of life survey form means of the this is a non-specific questionnaire for assessing the patient's quality of life.When 1 point-is the highest result (best),5 points-this is the lowest result (worst).
Change in frequency of involuntary urination (urinary incontinence) from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  The effectiveness was assessed using ICIQ-SF (International Urine Retention Index), a subjective indicator of the severity of urine loss and quality of life in patients with urinary incontinence, using the format of questions on a 5-point Likert scale to assess the presence, severity and concomitant symptoms. This is a subjective indicator designed to assess the level, impact and suspected cause of urinary incontinence on the quality of life.5 points-the highest score of the result,0 point- the lowest score of the result.The total amount of points for answering the questions where 0 points - a slight degree of urinary incontinence,19 - 21 - very severe urinary incontinence.
Change in frequency of involuntary urination during physical activities (stress urinary incontinence). | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the PISQ12 is a specific and reliable questionnaire consisting of three sections: behavioral and emotional characteristics, physical aspects and questions concerning the patient's relationship with a partner.Each item of the questionnaire contains five possible answers,which are evaluated in points.The result of the survey is expressed by the sum of points on all points.The maximum number of points is48,which is an indicator of the best sexual function. SF36 quality of life survey form means of the this is a non-specific questionnaire for assessing the patient's quality of life.When 1 point-is the highest result (best),5 points-this is the lowest result (worst)

SECONDARY OUTCOMES:
Change in burning pain in the vagina from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the Female Sexual Function Index (FSFI)- a self-controlled questionnaire survey, including 19 items,allows you to evaluate the features of desire,arousal,arousal,orgasm,achieving sexual satisfaction,and the presence of dyspareunia.With the help of this questionnaire,it is possible to conduct a differential assessment of clinical manifestations of sexual disorders.5 points-the highest score of the result,1 point- the lowest score of the result.

OTHER OUTCOMES:
Change in dyspareunia (discomfort during sexual intercourse) from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the Female Sexual Function Index (FSFI)- a self-controlled questionnaire survey, including 19 items,allows you to evaluate the features of desire,arousal,arousal,orgasm,achieving sexual satisfaction,and the presence of dyspareunia.With the help of this questionnaire,it is possible to conduct a differential assessment of clinical manifestations of sexual disorders.5 points-the highest score of the result,1 point- the lowest score of the result.
Change in frequency of sexual activity sensations during sexual intercourse (sensitivity and arousal) from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the Female Sexual Function Index (FSFI)- a self-controlled questionnaire survey, including 19 items,allows you to evaluate the features of desire,arousal,arousal,orgasm,achieving sexual satisfaction,and the presence of dyspareunia.With the help of this questionnaire,it is possible to conduct a differential assessment of clinical manifestations of sexual disorders.5 points-the highest score of the result,1 point- the lowest score of the result.
Change in satisfaction with sex life from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the Female Sexual Function Index (FSFI)- a self-controlled questionnaire survey, including 19 items,allows you to evaluate the features of desire,arousal,arousal,orgasm,achieving sexual satisfaction,and the presence of dyspareunia.With the help of this questionnaire,it is possible to conduct a differential assessment of clinical manifestations of sexual disorders.5 points-the highest score of the result,1 point- the lowest score of the result.
Change in frequency of orgasms during sexual intercourse from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by means of the Female Sexual Function Index (FSFI)- a self-controlled questionnaire survey, including 19 items,allows you to evaluate the features of desire,arousal,arousal,orgasm,achieving sexual satisfaction,and the presence of dyspareunia.With the help of this questionnaire,it is possible to conduct a differential assessment of clinical manifestations of sexual disorders.5 points-the highest score of the result,1 point- the lowest score of the result.
Change in general health condition from baseline | Questioning was conducted at the following time points: before laser treatment, one month after each laser treatment session, and 6 months after the last procedure.
  Efficacy was assessed by SF36 quality of life survey form means of the this is a non-specific questionnaire for assessing the patient's quality of life.When 1 point-is the highest result (best),5 points-this is the lowest result (worst) Calculations were made using the Subjective assessment questionnaire on a 10-point scale. Which included questions from each questionnaire:Female Sexual Function Index (FSFI),ICIQ-SF (International Urinary Continence Index), PISQ-12 survey form, SF36 quality of life survey form.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Budgetary Healthcare Institution "Volga District Medical Center" of the Federal Medical and Biological Agency, Nizhny Novgorod, Russia,Nighegorodskaya Oblast', Russia

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol,Statistical Analysis Plan (SAP).
Supporting Information: Study Protocol, SAP
Time Frame: The data can be viewed from the moment of registration of the clinical trial until December 2022.
Access Criteria: We provide access to data on request via email